CLINICAL TRIAL: NCT04539431
Title: Sensitive Diagnosis, Prognosis and Treatment Planning on Open Platform of Glioma Brain Tumours - E12513 - SensiScreen Glioma
Brief Title: Glioma Brain Tumours - E12513 - SensiScreen Glioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Collaborators: Istituto Cantonale di Patologia (Other); Neurocenter of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Milo Frattini, Head, Molecular Pathology Service, Ente Ospedaliero Cantonale, Bellinzona
Other Study IDs: ICP_glioma_001
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liquid biopsies, tissue block, blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: The cases with glioma will be identified in the databases of hospital, the material will be preliminarily evaluated in order to see if there is sufficient tissue left for analysis.
  Interventions: Genetic: validation of new technologies
- Prospective: A blood sample for molecular analyses will be collected in all the cases, CSF samples will be taken only if recommended by the normal surgical routine.
  Interventions: Genetic: validation of new technologies

INTERVENTIONS:
Genetic: validation of new technologies — Development of a new molecular assay on tissue as well as on liquid biopsies (plasma and CSF), based on a single, open, real-time PCR platform with unprecedented sensitivity

SUMMARY:
Validation of a new platform for the molecular characterization of patients affected by glioma. The new platform includes a series of faster, less expensive real-time PCR methodologies that, in comparison to standard analyses (DS, MS-PCR), are also characterized by higher sensitivity and consequently can be able to identify mutations in ctDNA extracted from liquid biopsies as well. The development of these assays will allow the analysis of molecular markers alteration even in liquid biopsies, providing a less invasive sampling than tissue biopsies, a procedure that sometimes is characterized by side effects or that allow the collection of few tissues for the histological and molecular diagnosis.

This study will not interfere with the patients routine treatment pathway and there will be no deviation from the standard of care: the molecular characterization of the tissues will be performed according to the standard diagnostic routine using the currently approved methodologies. For the retrospective study, it will be used the left-over DNA. For the cohort, that includes the collection and the subsequent analysis of liquid biopsies (prospective study), blood and CSF will be sampled during surgery.

The mutations in the molecular markers will be analyzed in tissue as well as in plasma and CFS samples by the new real-time based assays. Then, the qualitative and quantitative values obtained on liquid biopsies with the new methodology will be compared to the results of the standard methodologies already obtained, for diagnostic routine, on surgical tissue samples of the same patients.

ELIGIBILITY:
Retrospective Cohort

Inclusion Criteria:

* Patient with available tissue material or with available molecular data concerning the tissue biopsy obtained during surgery and analyzed for diagnosis

Exclusion Criteria:

* Insufficient amount of tumor cells in the tissue biopsy for the molecular characterization
* Inability to consent and follow the procedures of the study (for alive patients)

Prospective Cohort

Inclusion Criteria:

* Age ≥ 18 years old
* Affected by suspected glioma and requiring surgery
* Patient with available tissue material or with available molecular data concerning the tissue biopsy obtained during surgery and analyzed for diagnosis
* Written informed consent

Exclusion Criteria:

* Insufficient amount of tumor cells in the tissue biopsy for the molecular characterization
* Inability to consent and follow the procedures of the study
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by suspected glioma
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Demonstration that the new methodology improves the features | 2 hours
  Demostrate that are found at least the same number of mutations in comparison with respect to standard tests

CONTACTS AND LOCATIONS:
Overall Officials: Milo Frattini, PhD, Study Chair — Institute of Pathology
Locations (1):
- Institute of Pathology Ente Ospedaliero Cantonale, Locarno, Switzerland

IPD SHARING:
Plan to Share IPD: No